CLINICAL TRIAL: NCT03112473
Title: A Randomized, Controlled Clinical Trial of Upper Limb Training With Bilateral Cutaneous Electrical Stimulation to Improve Upper Limb Functions in Patients With Chronic Stroke
Brief Title: Effect of Bilateral TENS With TOT on Upper Limb Function in Patients With Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HMRF_SNg
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Results first posted 2021-04-20 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Stroke
Keywords: upper limb; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Stroke | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant and outcome assessor were blinded to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Bilateral TENS (Bi-TENS) group (Active Comparator): All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with bilateral electrical stimulation
  Interventions: Behavioral: Task-orientated training; Device: Transcutaneous electrical nerve stimulation (TENS)
- Unilateral TENS (uni-TENS) group (Placebo Comparator): All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with unilateral electrical stimulation on paretic side and sham electrical stimulation on the non-paretic side
  Interventions: Behavioral: Task-orientated training; Device: Transcutaneous electrical nerve stimulation (TENS); Device: Sham electrical nerve stimulation
- Placebo group (Placebo Comparator): All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with bilateral sham electrical stimulation
  Interventions: Behavioral: Task-orientated training; Device: Sham electrical nerve stimulation
- Control group (No Intervention): No Active intervention

INTERVENTIONS:
Behavioral: Task-orientated training — Task-Oriented Training (TOT) is a goal-directed exercise therapy, which help the people derive optimal control strategies for solving specific motor problems in real environment. In this study, TOT included stretching exercises, mobilizing exercise, strengthening exercises, seated reaching tasks, dexterity training and bimanual practice.
  Arms: Bilateral TENS (Bi-TENS) group; Placebo group; Unilateral TENS (uni-TENS) group
Device: Transcutaneous electrical nerve stimulation (TENS) — The stimulator was 120z Dual-Channel TENS Unit (ITO PHYSITHERAPY&REHABILITION CO., LTD, Tokyo, Japan). The parameter (100 Hz, 0.2 ms square pulses, intensity barely below the motor threshold) of TENS followed our previous study
  Arms: Bilateral TENS (Bi-TENS) group; Unilateral TENS (uni-TENS) group
Device: Sham electrical nerve stimulation — A identical-looking TENS devices that electrical circuit has been disconnected.
  Arms: Placebo group; Unilateral TENS (uni-TENS) group

SUMMARY:
On the basis that the combined use of Uni-TENS and TRT is an effective intervention in upper limb recovery, and the advantage of Bi-TENS eliciting extra neural pathway in the intact hemisphere to facilitate the motor recovery, There is a research gap in whether the Bi-TENS over both the paretic and non-paretic limbs could probably augment the treatment effects of TOT in upper limb motor control in people with stroke.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether Bi-TENS+TOT was superior to Uni-TENS+TOT, Placebo-TENS+TOT alone and no active treatment in improving the upper limb motor control and upper limb function and community integration in people with chronic stroke.

The null hypothesis will be that Bi-TENS+TOT is not significantly different from Uni-TENS+TOT,Placebo-TENS+TOT alone and no active treatment in improving the upper limb motor control and upper limb function and community integration in people with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be recruited from local self-help groups through poster advertising.
* Subjects will be included if they are between 50 and 80 years of age
* Have been diagnosed with ischaemic brain injury or intracerebral hemorrhage by MRI or computed tomography within the previous 1 to 10 years
* have volitional control of the non-paretic arm and at least minimal antigravity movement in the shoulder of the paretic arm,
* have at least 5º in wrist extension in the antigravity position,
* score > 6 out of 10 in the Abbreviated Mental Test, and
* are able to follow instructions and give informed consent.

Exclusion Criteria:

* • have any additional medical, cardiovascular or orthopedic condition

  * use a cardiac pacemaker
  * have receptive dysphasia
  * have a significant upper limb peripheral neuropathy
  * are involved in drug studies or other clinical trials, or
  * have severe shoulder, elbow, wrist or finger contractures that would preclude a passive range of motions of the arm, and
  * have a skin allergy that would prevent electrical stimulation.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-11-24 (Actual); Primary Completion 2020-10-24 (Actual); Study Completion 2020-10-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen P, Liu TW, Kwong PWH, Lai CKY, Chung RCK, Tsoh J, Ng SSM. Bilateral Transcutaneous Electrical Nerve Stimulation Improves Upper Limb Motor Recovery in Stroke: A Randomized Controlled Trial. Stroke. 2022 Apr;53(4):1134-1140. doi: 10.1161/STROKEAHA.121.036895. Epub 2021 Dec 2. PMID 34852645

RESULTS

PARTICIPANT FLOW:
Groups:
- Bilateral TENS (Bi-TENS) Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with bilateral electrical stimulation
  Task-orientated training: Bi/Uni/Placebo TENS and Task-orientated training on upper limb
  Transcutaneous electrical nerve stimulation (TENS)
- Unilateral TENS (Uni-TENS) Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with unilateral electrical stimulation on paretic side
  Task-orientated training: Bi/Uni/Placebo TENS and Task-orientated training on upper limb
  Transcutaneous electrical nerve stimulation (TENS)
- Placebo Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with bilateral sham electrical stimulation
  Task-orientated training: Bi/Uni/Placebo TENS and Task-orientated training on upper limb
  Sham electrical nerve stimulation
Period: Overall Study
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Started | 30 | 30 | 30 | 30
Completed | 30 | 30 | 30 | 30
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bilateral TENS (Bi-TENS) Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 7 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with bilateral electrical stimulation
- Unilateral TENS (Uni-TENS) Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 7 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with unilateral electrical stimulation on paretic side
- Placebo Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 7 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with bilateral sham electrical stimulation
- Total: Total of all reporting groups
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 21 | 23 | 22 | 89
  >=65 years | 7 | 9 | 7 | 8 | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.37 (7.13) | 62.30 (7.30) | 61.70 (6.70) | 61.70 (5.91) | 61.52 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 9 | 10 | 44
  Male | 18 | 17 | 21 | 20 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 30 | 30 | 30 | 30 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Hong Kong | 30 | 30 | 30 | 30 | 120
Fugl-Meyer Assessment of Upper Extremity [Mean (Standard Deviation); unit: units on a scale] — FMA-UE was used for evaluating the upper limb motor control from proximal to distal part of the limb, and voluntary movement from synergistic to isolated in people with stroke. The FMA-UE has shoulder-arm, wrist, hand and coordination and speed subsections. The score of shoulder-arm, wrist, hand and coordination and speed sub-scale are combined to compute the total score. The maximum total score is 66, with 33 items and ordinal scoring from 0 to 2. A higher score of FMA-UE indicated a higher level of upper limb motor control.
  units on a scale | 37.03 (12.02) | 41.83 (17.12) | 38.77 (15.78) | 43.93 (18.74) | 40.39 (16.13)

OUTCOME MEASURES:

1. Primary Outcome: Fugl Meyer Assessment on Upper Extremity (FMA-UE)
Description: FMA-UE was used for evaluating the upper limb motor control from proximal to distal part of the limb, and voluntary movement from synergistic to isolated in people with stroke. The FMA-UE has shoulder-arm, wrist, hand and coordination and speed subsections. The score of shoulder-arm, wrist, hand and coordination and speed sub-scale are combined to compute the total score. The maximum total score is 66, with 33 items and ordinal scoring from 0 to 2. A higher score of FMA-UE indicated a higher level of upper limb motor control.
Time Frame: Pre-intervention, Mid-intervention (4 weeks), Post-intervention (8 weeks), Follow-up 1 month (12 weeks), Follow-up 3 months (20 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Unilateral TENS (Uni-TENS) Group: All subjects will undergo 20 sessions of their assigned intervention (60 minutes, thrice a week, for 8 weeks). All subjects will receive 60 minutes task-oriented upper limb training (TOT) with unilateral electrical stimulation on paretic side
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale
  Pre-intervention | 37.03 (12.02) | 41.83 (17.12) | 38.77 (15.78) | 43.93 (18.74)
  Mid-intervention | 41.27 (13.38) | 43.60 (17.21) | 40.13 (15.41) | 44.87 (17.25)
  Post-intervention | 43.43 (13.73) | 44.23 (16.12) | 40.23 (14.97) | 44.20 (18.16)
  1-month followed up | 42.60 (13.36) | 42.70 (17.35) | 40.90 (14.43) | 45.03 (17.99)
  3-month followed up | 43.17 (13.61) | 43.17 (18.65) | 40.60 (14.67) | 45.23 (17.77)

2. Secondary Outcome: Jacket Test (JT)
Description: Jacket Test is one of the items in the Physical Performance Test. The subject is required to don a jacket or a cardigan sweater such that it is straight on his or her shoulders, and then remove it completely. The time for completing the task is recorded.(Rueben DB et al, 1990) This Jacket Test (JT) can be used to evaluate the functional mobility of the upper limbs as the test involves abduction of the shoulder joint, flexion and extension of the elbow joint and gripping with the hands.
Time Frame: as for outcome 1
Population: Nine subjects (Uni-TENS+TOT: 3; Placebo-TENS+TOT: 1; Control: 5) could not complete JT due to difficulty in maintaining the standing position without physical aids.
Measure: Mean (Standard Deviation); unit: second
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 27 | 29 | 25
second
  Pre-intervention | 36.51 (12.44) | 36.98 (22.02) | 36.87 (17.53) | 33.36 (21.39)
  Mid-intervention | 33.02 (13.66) | 35.78 (20.92) | 36.86 (15.53) | 32.58 (23.41)
  Post-intervention | 32.55 (11.70) | 30.67 (15.66) | 34.71 (16.08) | 34.08 (23.55)
  1-month followed-up | 33.35 (12.46) | 32.83 (20.32) | 34.24 (18.25) | 31.47 (21.79)
  3-month followed-up | 32.00 (12.51) | 32.54 (18.11) | 34.24 (17.19) | 31.77 (22.19)

3. Secondary Outcome: Maximal Voluntary Contraction (MVC)-Peak Torque
Description: The force data would be recorded by the self-made load cell. And the mean value peak torque of the joint would be calculated by the force and the length from the wrist joint to the head of 3rd metacarpal.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: N*m
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
N*m
  Peak Torque-wrist flexion-Pre-intervention | 3.69 (1.79) | 4.51 (2.63) | 4.86 (2.82) | 5.13 (2.29)
  Peak Torque-wrist flexion-Mid-intervention | 4.40 (1.90) | 4.77 (2.74) | 4.71 (2.74) | 5.35 (2.68)
  Peak Torque-wrist flexion-Post-intervention | 5.10 (2.17) | 4.74 (2.43) | 4.94 (2.58) | 5.39 (2.64)
  Peak Torque-wrist flexion- 1-month followed up | 4.86 (2.30) | 4.85 (2.60) | 5.17 (2.84) | 5.57 (2.72)
  Peak Torque-wrist flexion- 3-month followed up | 5.08 (2.12) | 4.89 (2.50) | 5.28 (2.62) | 5.70 (2.78)
  Peak Torque-wrist extension-Pre-intervention | 3.38 (1.95) | 3.12 (2.36) | 3.40 (2.17) | 3.64 (2.64)
  Peak Torque-wrist extension-Mid-intervention | 3.62 (1.70) | 3.10 (2.46) | 3.41 (2.48) | 3.55 (2.53)
  Peak Torque-wrist extension-Post-intervention | 3.77 (1.70) | 3.58 (2.74) | 3.81 (2.62) | 3.71 (2.39)
  Peak Torque-wrist extension- 1-month followed up | 3.87 (1.89) | 3.67 (2.82) | 3.61 (2.35) | 3.81 (2.34)
  Peak Torque-wrist extension- 3-month followed | 3.91 (1.98) | 3.86 (2.76) | 3.66 (2.86) | 3.98 (2.67)

4. Secondary Outcome: Action Research Arm Test (ARAT)
Description: ARAT will be used to assess the 4 aspects of upper limb function(grasp, grip, pinch and gross arm movement). This scale is consistent of 19 items. The quality of performance on each item is rated from 0-3, so the score of ARAT is ranged from 0-57. The score of rasp, grip, pinch and gross arm movement sub-scale are combined to compute the total score. The scores for the 15 tasks will be summed and then averaged to yield the mean functional ability score. A higher ARAT score indicated a higher upper limb motor function.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale
  Pre-intervention | 28.70 (20.09) | 31.73 (20.09) | 28.30 (21.69) | 34.97 (21.97)
  Mid-intervention | 31.27 (20.86) | 33.93 (20.27) | 29.40 (20.85) | 35.30 (21.61)
  Post-intervention | 33.40 (19.77) | 33.13 (20.80) | 30.30 (21.65) | 36.07 (22.85)
  1-month followed-up | 31.33 (19.24) | 34.90 (19.74) | 31.03 (21.83) | 36.77 (21.79)
  3-month followed-up | 32.20 (20.12) | 33.33 (21.17) | 30.43 (21.97) | 36.27 (22.29)

5. Secondary Outcome: The Range of Motion (ROM) of Upper Limb Joints
Description: With 0° shoulder flexion and 90° elbow flexion, the forearm and wrist will be placed in a neutral position in the relaxed phase. When the task begins, the subjects will be asked to perform the full range of motion for wrist flexion/extension. With 90° shoulder flexion and 0° elbow flexion, the forearm will be placed in a neutral position in the relaxed phase. When the task begins, the subjects will be asked to perform the full range of motion for elbow flexion/extension.
  All the subjects will be requested to perform their joint ROM to the best of their abilities.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: degree
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
degree
  Elbow-Pre | 76.67 (28.89) | 85.73 (27.30) | 82.88 (24.01) | 90.22 (33.36)
  Elbow-Mid | 84.70 (22.96) | 84.33 (28.58) | 86.75 (22.64) | 79.28 (29.33)
  Elbow-Post | 87.70 (23.78) | 88.47 (26.07) | 83.60 (18.82) | 86.75 (23.06)
  Elbow-1-month followed-up | 84.13 (30.91) | 84.05 (29.51) | 81.85 (23.81) | 89.67 (26.64)
  Elbow-3-month followed-up | 85.13 (33.79) | 89.90 (30.74) | 81.95 (20.10) | 87.02 (27.53)
  Wrist-Pre | 72.42 (40.84) | 69.97 (49.52) | 72.70 (44.04) | 87.41 (48.28)
  Wrist-Mid | 71.43 (36.45) | 74.77 (47.35) | 62.23 (50.02) | 87.72 (40.34)
  Wrist-Post | 73.83 (35.51) | 75.42 (47.96) | 69.77 (42.35) | 90.07 (42.02)
  Wrist-1-month followed-up | 72.92 (37.84) | 78.30 (48.23) | 66.05 (38.46) | 87.97 (46.11)
  Wrist-3-month followed-up | 70.67 (39.57) | 78.32 (54.34) | 71.18 (44.39) | 90.78 (45.25)

6. Secondary Outcome: Motor Activity Log (MAL)
Description: The MAL questionnaire will be used to assess how frequently and how well a person uses the paretic upper limb in 30 activities of daily life in a semi-structured interview. Based on a six-point ordinal scale, subjects will be required to rate (1) the amount of use (AOU), and (2) the quality of movement (QOM) when performing these 30 tasks in real life situations. Each task was rated from 0 to 5. The score of the 30 activities of daily life were combined to compute the total score of MAL-AOU and MAL-QOM, respectively. Hence, the total score of AOU and QOM component were rated from 0 to 150. The higher MAL-AOU score indicated a higher frequency use of the paretic upper limb, and the higher MAL-QOM score indicated a higher movement quality of the paretic upper limb.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale
  AOU-Pre | 34.03 (30.35) | 49.72 (47.73) | 39.20 (40.54) | 45.28 (34.50)
  AOU-Mid | 35.57 (35.59) | 44.93 (47.92) | 53.27 (50.99) | 47.73 (43.91)
  AOU-Post | 38.53 (38.86) | 48.87 (49.56) | 54.70 (50.15) | 45.10 (44.62)
  AOU-1-month followed-up | 35.95 (31.91) | 48.68 (49.49) | 48.58 (50.04) | 49.25 (50.86)
  AOU-3-month followed-up | 39.80 (34.42) | 58.03 (54.14) | 50.53 (48.84) | 46.42 (46.33)
  QOM-Pre | 42.10 (36.15) | 56.92 (49.89) | 52.42 (45.09) | 58.00 (43.44)
  QOM-Mid | 41.83 (37.57) | 53.20 (47.32) | 61.10 (53.46) | 51.53 (46.79)
  QOM-Post | 40.93 (35.97) | 61.38 (53.73) | 51.53 (46.76) | 52.77 (44.83)
  QOM-1-month followed-up | 43.05 (35.85) | 54.00 (51.32) | 54.88 (53.83) | 57.13 (53.52)
  QOM-3-month followed-up | 43.28 (39.07) | 59.08 (54.20) | 54.23 (50.13) | 57.18 (50.78)

7. Secondary Outcome: Chinese Version of Community Integration Measure (CIM)
Description: The Chinese version of CIM was used to assess the level of community integration of the subjects. The CIM-C has been shown to have good internal consistency and good test-retest reliability for people with stroke . CIM has 10 items, each item rate from 1-5, giving a minimum score of 10 to a maximum of 50. A higher score indicated a higher level of community integration.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
score on a scale
  Pre-intervention | 39.47 (7.51) | 41.23 (6.89) | 41.87 (8.02) | 39.67 (9.21)
  Mid-intervention | 41.23 (6.60) | 39.90 (11.79) | 42.20 (7.40) | 38.37 (9.04)
  Post-intervention | 40.17 (7.04) | 41.67 (9.66) | 42.17 (8.33) | 39.80 (9.31)
  1-month followed-up | 41.63 (6.96) | 42.70 (12.92) | 43.17 (7.00) | 39.33 (9.08)
  3-month followed-up | 40.10 (7.16) | 40.23 (10.45) | 41.03 (7.93) | 41.10 (8.86)

8. Secondary Outcome: Maximal Voluntary Contraction (MVC)-Cocontraction Ratio
Description: EMG signal of Radial Carpi Extensor and Ulnar Carpi Flexor for both affected and unaffected side would be recorded by the surface EMG electrodes when asked the subjects to perform the MVC of wrist extension and flexion for 5s in each trial. Each movement would perform 3 times. The data of the 3 trials will be averaged. The co-contraction ratio would be calculated by the iEMG area of antagonist to total (agonist+antagonist), which would be captured for 0.5s from the window began at 0.25s before and ended at 0.25s after the peak value of MVC.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
Number analyzed (Participants) | 30 | 30 | 30 | 30
ratio
  Co-contraction Ratio of Wrist Flexion-pre | 0.28 (0.14) | 0.24 (0.11) | 0.25 (0.15) | 0.24 (0.13)
  Co-contraction Ratio of Wrist Flexion-mid | 0.26 (0.13) | 0.27 (0.13) | 0.23 (0.11) | 0.24 (0.13)
  Co-contraction Ratio of Wrist Flexion-post | 0.26 (0.14) | 0.28 (0.12) | 0.25 (0.12) | 0.24 (0.12)
  Co-contraction Ratio of Wrist Flexion-follow up 1 month | 0.26 (0.16) | 0.26 (0.11) | 0.25 (0.10) | 0.25 (0.13)
  Co-contraction Ratio of Wrist Flexion-follow up 3 months | 0.27 (0.16) | 0.25 (0.11) | 0.23 (0.15) | 0.23 (0.11)
  Co-contraction Ratio of Wrist Extension-pre | 0.29 (0.16) | 0.31 (0.23) | 0.25 (0.15) | 0.23 (0.18)
  Co-contraction Ratio of Wrist Extension-mid | 0.25 (0.12) | 0.28 (0.20) | 0.26 (0.15) | 0.22 (0.18)
  Co-contraction Ratio of Wrist Extension-post | 0.27 (0.14) | 0.28 (0.21) | 0.28 (0.16) | 0.27 (0.20)
  Co-contraction Ratio of Wrist Extension-follow up 1 month | 0.29 (0.17) | 0.28 (0.23) | 0.26 (0.14) | 0.23 (0.15)
  Co-contraction Ratio of Wrist Extension-follow up 3 months | 0.28 (0.18) | 0.27 (0.18) | 0.27 (0.15) | 0.22 (0.14)

ADVERSE EVENTS:
Time Frame: 5 months (from the baseline to the follow up 3 months assessment)
Description: Baseline: There was no adverse event occurred in baseline, Mid-Intervention, Post-intervention, follow-up 1 month and follow-up 3 month.
Arm/Group | Bilateral TENS (Bi-TENS) Group | Unilateral TENS (Uni-TENS) Group | Placebo Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
1. The time window of the assessment may not be widen enough to observe the change in all the outcomes.
2. The sample size may not be large enough provide sufficient power to detect the improvement in all the outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-03-01): https://cdn.clinicaltrials.gov/large-docs/73/NCT03112473/Prot_SAP_ICF_000.pdf